CLINICAL TRIAL: NCT03946579
Title: Evaluation of the Quality of Life and Sexuality of Patients Over 65 Years of Age Undergoing Adjuvant Treatment for Breast Cancer
Brief Title: Quality of Life and Sexuality of Patients Over 65 Years Undergoing Adjuvant Treatment for Breast Cancer
Acronym: QUALITY-AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB18.04
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: sexual health; quality of life; adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient treated by adjuvant therapy (Other): Self questionnaires of sexual health and quality of life (FSFI, QLQ-C30, BR23, ELD 15, HADS, GDS 15, BIS, FACIT)
  Interventions: Other: self questionnaires

INTERVENTIONS:
Other: self questionnaires — FSFI, QLQ-C30, BR23, ELD15, HADS, GDS 15, FACIT, BIS

SUMMARY:
The purpose of this study is to assess the quality of life and sexuality during adjuvant chemotherapy in over 65 years old patients with breast cancer

DETAILED DESCRIPTION:
Evaluation of quality of life and sexual health will be assessed by the mean of validated self questionnaires after surgery for breast cancer, before and after adjuvant chemotherapy and one year after initial surgery

ELIGIBILITY:
Inclusion Criteria:

* Women over 65 years of age
* treatment by adjuvant therapy for breast cancer
* pTxNxM0
* sexually active at least three months before inclusion
* in couple or not

Exclusion Criteria:

* Inflammatory breast cancer
* Not sexually active before breast cancer diagnosis
* Opposition to fill sel questionnaire and collection of the data

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Assessment of Sexual Health | one year
  assessment with Female sexual functionnal index (FSFI) self questionnaire

SECONDARY OUTCOMES:
Assessment of Quality of life | one year
  assessment with the Quality of life questionnaire (QLQ-C30) that contains 30 items dealing with fatigue, pain, nausea and vomiting, general condition and social, emotional and cognitive functions.
Assessment of Body Image | one year
  assessment with body image scale that contains 10 items dealing with body image
Assessment ofTiredness | one year
  assessment with Functionnal assessment of chronic illness therapy-Fatigue (FACIT-F) self questionnaire that contains 13 items dealing with fatigue
Assessment of Anxiety | one year
  assessment with Hospital anxiety and depression scale (HADS) that contains 15 items dealing with anxiety
Assessment of Depression | one year
  assessment geriatric depression scale (GDS 15 self questionnaire) that contains 15 item dealing with depression

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rigal, MD, Principal Investigator — Centre Henri Becquerel
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - Centre François Baclesse, Caen
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No